CLINICAL TRIAL: NCT05934123
Title: Effects of Implementation of a Care Bundle on Rates of Necrotising Enterocolitis and Own Mother's Milk Feeding in the East Midlands: a Mixed Methods Impact and Process Evaluation Study
Brief Title: Effects of Implementation of a Care Bundle on Rates of NEC and Own Mother's Milk Feeding in the East Midlands
Acronym: EMNODN-NEC
Status: Completed | Type: Observational
Sponsor: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Collaborators: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: UHDB/2021/059
Record Dates: First submitted 2023-03-23; First posted 2023-07-06 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-02

CONDITIONS: Necrotising Enterocolitis Neonatal
Keywords: Breastfeeding; Necrotising enterocolitis; Care bundle
MeSH Terms: conditions — Enterocolitis, Necrotizing; Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Intervention group: Infants admitted to the 11 EMNODN neonatal units
  Interventions: Behavioral: EMNODN NEC Care Bundle

INTERVENTIONS:
Behavioral: EMNODN NEC Care Bundle — A care bundle created by the East Midlands Neonatal Operational Delivery Network to guide neonatal services in the region to implement practices that support own mother's milk feeding and other interventions that may reduce the risk of NEC in babies born <32 weeks' gestational age.

SUMMARY:
Necrotising enterocolitis (NEC) is a life-threatening gut disease in babies born early. Feeding preterm babies their own mother's milk prevents NEC. Fewer babies in the East Midlands get their own mother's milk than the national average, and more babies get NEC.

The East Midlands Neonatal Operational Delivery Network (EMNODN) has created a care bundle to increase own mothers' milk feeding and reduce rates of NEC among babies born more than 8 weeks early, who are at the greatest risk of NEC. The care bundle describes the support that parents can expect to receive to help mothers feed their breastmilk to their babies. It also provides guidelines to help neonatal units ensure babies receive optimum nutritional care.

This study will find whether this bundle is effective in helping more babies receive their own mothers' milk and in reducing NEC. It will also identify how well the bundle was introduced and which parts of the bundle were most helpful.

The study team will answer these questions by collecting and studying data from babies' medical records.

DETAILED DESCRIPTION:
Necrotising enterocolitis (NEC) is a serious, life-threatening disease in preterm infants. Preterm birth, affecting over 52,000 babies per year (around 7.3% of live births), is the largest cause of neonatal mortality in the UK. The 2019 NHS Long Term Plan aims to reduce neonatal mortality by 50% with plans to "improve the safety and effectiveness of neonatal critical care" and "enhance the experiences of families" during this worrying period.

An estimated 12% of infants born weighing <1500g develop NEC and 30% of these die. Survivors have an increased risk of adverse neurodevelopmental outcomes, including cerebral palsy and cognitive impairment. In the UK, NEC rates are collected by the National Neonatal Audit Programme (NNAP), a national audit run by the Royal College of Paediatrics and Child Health, commissioned by the Healthcare Quality Improvement Partnership (https://nnap.rcpch.ac.uk).

The East Midlands Neonatal Operational Delivery Network (EMNODN) (https://www.emnodn.nhs.uk) is one of 11 clinically managed Neonatal Operational Delivery Networks in England. ODNs were formed, in 2003, by the Department of Health, to ensure that babies and their families receive high quality, equitable and accessible care. The rate of NEC in the EMNODN has remained above the national average since 2017 (when this measure was added to NNAP) and there are wide variations between units.

Preterm infants are unable to directly suckle on the breast. Mothers express breastmilk which is fed to their infant via an oro/nasogastric tube. As infants grow and mature, they develop the ability to suck and swallow and establish breastfeeding. Some infants continue to receive own mother's milk via a cup, syringe, or bottle as per parental choice; all these are included within 'own mother's milk feeding'. Encouraging and supporting own mother's milk feeding prevents NEC and has several additional advantages, including improved long-term neurodevelopment and parent-infant bonding. Health economic analysis estimates that if all premature infants were fed own mother's milk, the total lifetime cost saving to the NHS would be £46.7 million (£30.1 million in the first year of life) and there would be 238 fewer deaths per year with a gain of £153.4 million in lifetime productivity. The adjusted incremental costs of medical NEC and surgical NEC over and above the average costs incurred for extremely premature infants without NEC, in 2011, were estimated to be $74,004 (95% confidence interval (CI), $47,051-$100,957) and $198,040 (95% CI, $159,261-$236,819) per infant, respectively.

Early start and continuation of feeding with own mother's milk, such that babies go home breastfeeding, is vital to ensure babies continue to receive own mother's milk throughout neonatal care and remain at a reduced risk of NEC. Unfortunately, in NNAP, rates of any breast milk feeding at discharge in EMNODN have been consistently below the national average, again with wide local variations.

National recommendations cite a need for quality improvement (QI) efforts to boost own mother's milk feeding to reduce NEC. In 2020, NNAP recommended that "if rates of NEC are relatively high, seek to identify and implement potentially better practices" and to "focus on the early initiation and sustainment of breastmilk feeding in conjunction with parents by reviewing data and processes" and "undertake selected QI activities suited to the local context". In keeping with this, the EMNODN has created a NEC Care Bundle which was introduced it to the 11 neonatal units in September 2022, with use fully embedded by December 2022.

Care bundles are a group of evidence-based interventions related to a disease or care process that, when executed together, result in better outcomes than when implemented individually. Interventions should be evidence-based, accepted as best practice, simple to implement, and part of day-to-day practice. This care bundle consists of recommendations, and parent-facing information, created by a multi-disciplinary team. It contains recommendations in two main areas: promotion of own mother's milk feeding and optimising nutritional care of preterm infants by ensuring early and adequate parenteral nutrition, given when infants cannot have sufficient milk feeds such as in the first hours after birth, while building milk feeds and when unwell, oropharyngeal colostrum (practice of giving own mothers' first milk directly into the infant's oropharynx to enhance immunity and protect against NEC), optimal time and speed of increasing milk feeds, and use of other interventions such as human donor milk, probiotics and breast milk fortifiers.

There is some evidence that QI programmes using care bundles can improve rates of own mother's milk feeding in neonatal units. A study in the East of England showed that introduction of a care bundle increased the prevalence of own mother's milk feeding from 50 to 57%. While such previous studies have looked at some measures of effectiveness of implementation, none have explored the effect of complex interventions on NEC rates and other feeding practices.

ELIGIBILITY:
Inclusion Criteria:

* All infants born at <32 weeks' gestational age admitted for neonatal care in England and Wales between 01/01/2016 to 30/09/2023 and who survived at least 48 hours

Exclusion criteria:

* Infants whose data are not included in the National Neonatal Research Database (NNRD)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include all infants born at <32 weeks gestational age who are admitted to a neonatal unit in England and Wales which contributes data to the National Neonatal Research Database (NNRD).
Sampling Method: Probability Sample
Enrollment: 53600 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Receiving any own mother's milk at discharge | Evaluation phase (01/23-09/23) compared to pre-implementation phase (01/16-08/22)
  Incidence rate ratio for incidence of receiving any own mother's milk at discharge in evaluation phase compared to pre-implementation phase
Receiving any own mother's milk on day 14 of life | Evaluation phase (01/23-09/23) compared to pre-implementation phase (01/16-08/22)
  Incidence rate ratio for incidence of receiving any own mother's milk on day 14 of life in evaluation phase compared to pre-implementation phase
Severe NEC requiring surgery or resulting in death | Evaluation phase (01/23-09/23) compared to pre-implementation phase (01/16-08/22)
  Incidence rate ratio for incidence of severe NEC requiring surgery or resulting in death in evaluation phase compared to pre-implementation phase

SECONDARY OUTCOMES:
Exclusive own mother's milk feeding at discharge | Evaluation phase (01/23-09/23) compared to pre-implementation phase (01/16-08/22)
  Incidence rate ratio for incidence of exclusive own mother's milk feeding at discharge in evaluation phase compared to pre-implementation phase
Any NEC, including NEC not requiring surgery and not resulting in death | Evaluation phase (01/23-09/23) compared to pre-implementation phase (01/16-08/22)
  Incidence rate ratio for incidence of any NEC in evaluation phase compared to pre-implementation phase

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Ojha, PhD, Principal Investigator — University of Nottingham
Locations (1):
- University Hospitals of Derby and Burton NHS Foundation Trust, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abramson J, Szatkowski L, Bains M, Orton E, Budge H, Spruce M, Ojha S. Effects of implementation of a care bundle on rates of necrotising enterocolitis and own mother's milk feeding in the East Midlands: protocol for a mixed methods impact and process evaluation study. BMJ Open. 2024 May 30;14(5):e078633. doi: 10.1136/bmjopen-2023-078633. PMID 38816042
- See also: Description of EMNODN Care Bundle — https://www.emnodn.nhs.uk/_files/ugd/143840_5050aa59d39b4c66bf2582d7491ba478.pdf